CLINICAL TRIAL: NCT05300425
Title: Leptospirosis, Tularaemia and Hepatitis E in a Rural Mountain Valley in the Alpine Region of Switzerland - A Cross-sectional Exploratory Seroprevalence Study
Brief Title: Seroprevalence of Leptospirosis in Val Müstair, Switzerland
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02409; am22Osthoff
Record Dates: First submitted 2022-03-16; First posted 2022-03-29 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Leptospirosis; Hepatitis E Virus Infection; Tularemia
Keywords: seroprevalence; Val Müstair Graubünden; Switzerland
MeSH Terms: conditions — Leptospirosis; Hepatitis E; Tularemia | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be stored at -20°C in a dedicated freezer, situated at the Hospital of Val Müstair and will be transferred to a dedicated at -80°C with limited access at the University Hospital Basel after recruitment is complete. If appropriate consent is granted, the samples not used in the study will be biobanked and may be used in future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample collection — Blood sample collection (at baseline and approximately two years after baseline). Enzyme-linked immunosorbent assays will be used to screen for IgG and IgM antibodies directed against the three pathogens (Leptospirosis, Tularemia, Hepatitis E).
Other: Data collection — Data collection on sociodemographic questions e.g. profession, leisure activities, animal contact

SUMMARY:
Human leptospirosis is a zoonotic disease caused by bacteria of the genus Leptospira. Due to its frequent inapparent course or mild severity with unspecific symptoms and limited availability of diagnostic laboratories the incidence of leptospirosis is likely to be underestimated. The hospital of Val Müstair is the major healthcare provider of a rural mountain valley in the canton of Graubünden/ Switzerland with approximately 1500 inhabitants. A relevant prevalence of Leptospira spp. antibodies in the population of the Val Müstair due to its geographic and social risk profile for Leptospira infection, namely the close contact of the population to both livestock and wildlife in agriculture and hunting is estimated. The aim of this study is to analyze the burden of this disease in order to evaluate the need of preventive measures. In addition, seroepidemiological data for the Hepatitis E virus (HEV) and for tularemia will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Aged 18 years or older
* Living for at least one year mainly (>6 months per year) in Val Müstair (including Taufers and Rifair, Italy)

Exclusion Criteria:

* Inability to give consent
* Inability to follow procedures
* Acute infections/inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 250 participants presenting to the medical office of the Hospital of Val Müstair will be included. There will be a consecutive ongoing recruitment through the medical staff in daily clinical practice and during regular blood donation days. Risk populations (hunters and farmes, national park rangers) will be directly addressed (newspaper announcement and via associations).
Sampling Method: Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Change in presence of antibodies against Leptospira spp, Francisella tularensis and Hepatitis E | at baseline and approximately two years after baseline (project duration for each patient is one day or two days respectively, if they agree for another blood sampling in two years)
  Change in presence of antibodies against Leptospira spp, Francisella tularensis and Hepatitis E evaluated by serology at two different time points

SECONDARY OUTCOMES:
Change in presence of antibodies in risk populations (hunters and farmers) | at baseline and approximately two years after baseline (project duration for each patient is one day or two days respectively, if they agree for another blood sampling in two years)
  Change in presence of antibodies against Leptospira spp., Hepatitis E and Francisella tularensis and of all pathogens in risk populations (hunters and farmers)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osthoff, PD Dr. med., Principal Investigator — University Hospital Basel, Division of Internal Medicine
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Division of Internal Medicine, Basel
  - Center da sanda Val Muestair, Val Müstair